CLINICAL TRIAL: NCT03500458
Title: Impact of Sleep Extension on Insulin Sensitivity and Dietary Intake in Adolescents
Brief Title: Impact of Sleep Extension in Adolescents
Acronym: SUNRISE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 17-2095; K23DK117021 (NIH); R03DK131225 (NIH)
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Insulin Sensitivity; Sleep; Dietary Habits
MeSH Terms: conditions — Insulin Resistance; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Typical Sleep (No Intervention): All participants will sleep for 6 nights (Sunday - Thursday) in the home environment per their usual school schedule.
- Sleep Extension (Experimental): Participants will be prescribed a sleep schedule that allows them to obtain 1 hour more time in bed compared to Typical Sleep. For participants completing the study September 2021 and later, they will also be instructed to take exogenous melatonin (500mcg) and maintain dim light conditions 2 hours before bedtime, and use light glasses for 30 minutes in an upright position after waking in the morning (Sleep Extension + Circadian Manipulation).
  Interventions: Behavioral: Sleep Extension

INTERVENTIONS:
Behavioral: Sleep Extension — Participants will be asked to increase time in bed at least 1 hour more than baseline
  Arms: Sleep Extension

SUMMARY:
Many teenagers do not get enough sleep. Obesity and diabetes are increasing in teenagers as well. This study plans to learn more about sleep and insulin resistance (insulin not working) in teenagers, and how these things may be related depending on sleep. This is important to know so that the investigators understand how sleep may play a role in health conditions like extra weight gain (increased food intake and less physical activity) and diabetes. To answer this question, the investigators plan to enroll teenagers who get <7 hours of sleep on school nights and measure changes in insulin sensitivity and dietary intake after a week of typical sleep (sleeping on their normal school schedule) and a week of longer sleep (spending 1+ hour longer in bed each night).

ELIGIBILITY:
Inclusion Criteria:

1. High school students between the age of 14-19 years
2. have typically insufficient sleep, defined by ≤ 7 hours per night on school days
3. BMI 5th-84th percentile for age and sex
4. habitually sedentary (< 3 hours of regular physical activity per week)
5. Tanner stage 4 or 5, based on breast development for girls and testicular size for boys.

Exclusion Criteria:

1. Any medications that affect IR or sleep (e.g., metformin, stimulants, atypical antipsychotics, current use of oral steroids)
2. regular use of melatonin or other sleep aids
3. a prior diagnosis of a sleep disorder (e.g. insomnia, delayed sleep phase syndrome, obstructive sleep apnea)
4. Type 2 diabetes or prediabetes
5. IQ<70 or severe mental illness that may impact sleep or ability to consent/assent (e.g., schizophrenia, psychotic episodes)
6. teens not enrolled in a traditional high school academic program (e.g., home school students)
7. schedules that would preclude participants from adhering to the sleep manipulation (e.g. night shift employment)
8. travel across more than two time zones in the 2 weeks prior to the study.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insulin Sensitivity | 2 weeks after Baseline and 7 weeks after Baseline
  Insulin sensitivity assessed two times with an insulin-modified intravenous glucose tolerance test.
Change in Sleep Duration & Timing | At Baseline, 1 week after Baseline, and 6 weeks after Baseline
  Assessed three times with a wrist-worn Actigraphy
Change in Physical activity | At Baseline, 1 week after Baseline and 6 weeks after Baseline
  Assessed three times with a triaxial thigh-worn ActivPal
Change in Dietary Intake | 1 week after Baseline and 6 weeks after Baseline
  Participants will be asked to complete diet diaries two times for 3 days during each sleep condition (prior to each overnight assessment), listing all food and drink consumed, estimated portion size, and timing of consumption.

SECONDARY OUTCOMES:
Change in glycemic variability | 2 weeks after Baseline and 7 weeks after Baseline
  Assessed two times with a continuous glucose monitor
MTNR1B rs10830963 SNP | 2 weeks after Baseline
  Genotyping will be conducted on saliva samples

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Simon, PhD, Principal Investigator — Children's Hospital Colorado and University of Colorado Anschutz Medical Campus
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No